CLINICAL TRIAL: NCT04941456
Title: Is Ambulation Distance on the Six-minute Walk Test Improved With the Use of Passy-Muir Valve for Patients With Tracheostomy Compared to Patients With an Open Tracheostomy?
Brief Title: Does Endurance Improve With the Use of Passy-Muir Valve for Patients With Tracheostomy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaylord Hospital, Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202104CUT
Record Dates: First submitted 2021-06-11; First posted 2021-06-28 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: PMV; Exercise Endurance; Tracheostomy
Keywords: Tracheostomy; PMV; Passy Muir Valve; Activity Tolerance; Intra-Thoracic Pressure; Six minute walk test; Borg Rating of Perceived Exertion; Oxygen Saturation

STUDY DESIGN:
Intervention Model Description: 6 period Quasi-Randomized Crossover Controlled Study. Enrollment will occur based off tracheostomy census report, site investigators will perform weekly pull of tracheostomy report to recruit appropriate patients.
Masking Description: Participants and care providers are unable to be masked to the intervention arm due to the nature of the study. As data was collected, investigators were unable to blind the data prior to exporting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Open Tracheostomy, Then Speaking Valve (Experimental): Participants perform the six-minute walk test each study session to assess ambulation distance, first using with an open tracheostomy on day 1 and then switching to a Passy-Muir Valve on day 2. Participants will alternate back and forth between open tracheostomy and Passy-Muir Valve until 3 sessions are completed with each condition.
  Interventions: Other: Open Tracheostomy; Device: PMV in place
- Speaking Valve, Then Open Tracheostomy (Experimental): Participants perform the six-minute walk test each study session to assess ambulation distance, first using the Passy-Muir Valve on day 1 and then switching to an open tracheostomy on day 2. Participants will alternate back and forth between the Passy-Muir Valve and open tracheostomy until 3 sessions are completed with each condition.
  Interventions: Other: Open Tracheostomy; Device: PMV in place

INTERVENTIONS:
Other: Open Tracheostomy — Participants will perform the six minute walk test with an open tracheostomy. Participants will complete 1 to 3 session over approximately three-weeks.
  Other Names: Standard
Device: PMV in place — Participants will perform the six minute walk test with a PMV in place. Participants will complete 1 to 3 sessions over approximately three-weeks.
  Other Names: PMV; Passy-Muir Valve

SUMMARY:
The purpose of this study is to determine if the use of the Passy-Muir Valve improves endurance for patients in the Long Term Acute Care setting as measured with the Six- Minute Walk Test.

DETAILED DESCRIPTION:
A Passy-Muir Valve (PMV) is a one-way valve that blocks air flow from exhalation in patients with a tracheostomy, and redirects it through to the upper airway to enable functional use of the glottis.

Typically, PMVs are used to assist patients being weaned from mechanical ventilation to communicate more effectively after tracheostomy. Devices are available that can be used in-line with the ventilator, as well as after ventilator liberation with a tracheostomy collar. PMVs provide patients with the ability to communicate, swallow, and improve diaphragmatic strength, which lengthens the periods of time that patients remain free from ventilator assistance, which ultimately leads to decannulation.

Use of the PMV during physical therapy helps restore the pressure support in the trunk, allowing for natural increases in intra-thoracic pressure (ITP) and intra-abdominal pressures (IAP) in response to increased postural demands. With an open tracheostomy tube and therefore, an open system, thoracic pressures cannot be increased or sustained as airflow passes through the tracheostomy tube and bypasses the upper airway. This difficulty would be observed when a patient needs to crawl, sit, push, or stand up. The typical means of gross motor movement for mobility is to engage the glottis (vocal cords) to restrict the expiratory lung volume in order to stabilize the chest and upper body. Placing a PMV on the tracheostomy tube closes the system and restores a patient's ability to use the upper airway to control expiratory flow and improve ITP and IAP.

The Six-Minute Walk Test (6MWT) is a commonly used test for the objective assessment of functional exercise capacity for management of patients with moderate to severe pulmonary disease. The patient is asked to walk as far as possible along a 30 meter minimally trafficked corridor for a period of six minutes. The 6MWT is a safe test with rare complications, the most common adverse event is oxygen desaturation below 80%.

Participants will consist of inpatients with tracheostomy who can tolerate use of Passy-Muir Valve; participants will be approached and consented into the study within 72 hours of being deemed medically appropriate for PMV use by medical staff. The 6MWT will be administered each session to assess ambulation distance, alternating open tracheostomy vs Passy-Muir Valve in place on sequential days to compare results. The Borg Rating of Perceived Exertion (RPE) scale will be administered before and after each session to assess patient's subjective rating of physical exertion levels on a scale from 6 through 20; 20 being the most exertion possible. Oxygen saturation and heart rate will be monitored before and after each session via pulse oximeter to assess for physiologic appropriateness of exercise response. For safety of the participant, while performing the six-minute walk test, participants will be allowed to use assistive devices as prescribed by the participant's primary physical therapist.

Sample size: A convenience sample of 30 participants will be collected.

Data: All data will be collected and analyzed in a paired fashion as appropriate; adjustments for abnormal distribution, unequal variance, and repeated measure will be applied as necessary. In the case of missing or inconsistent data due to early withdraw, early participant discharge, or other unforeseen events, the datasets will be evaluated as normal. Paired T-test and Repeated Measures Analysis of Variance (ANOVA) will be conducted to evaluate differences in Borg RPE scores and six-minute walk tests, between treatment arms, as appropriate. Correlation analysis may also be conducted to evaluate if there is any correlation to treatment arm, Borg RPE scores, six-minute walk test, and other variables such as session number.

ELIGIBILITY:
Inclusion Criteria:

1. Individual with tracheostomy who can tolerate daily 30 minute Physical Therapy sessions with use of PMV and be able to maintain oxygen saturations above 88% with exertion.
2. Ability to understand and respond to simple verbal instructions and one step commands in English well enough to consent without any interpretation.
3. Ability to ambulate a minimum of 10 feet with/without assistive device and with/without physical assistance.

Exclusion Criteria:

1. Active seizures
2. Active Pregnancy
3. Uncontrolled hypertension
4. Cognitive deficits that would disrupt ability to provide informed consent
5. Enteric infection control precautions
6. Ongoing orthostasis
7. Actively on decannulation protocol
8. Medical instability that would cause a doctor to put therapy program on hold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Cutler, DPT, Principal Investigator — Gaylord Hospital
Locations (1):
- Gaylord Hospital, Wallingford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Copies of the study protocol will be provided upon reasonable request. Requests for copies of deidentified study data will considered on a case by case basis.

REFERENCES:
- [Background] Massery M, Hagins M, Stafford R, Moerchen V, Hodges PW. Effect of airway control by glottal structures on postural stability. J Appl Physiol (1985). 2013 Aug 15;115(4):483-90. doi: 10.1152/japplphysiol.01226.2012. Epub 2013 Jun 13. PMID 23766504
- [Background] Roberts KJ. Enhancing Early Mobility With a Speaking Valve. Respir Care. 2020 Feb;65(2):269-270. doi: 10.4187/respcare.07671. No abstract available. PMID 31988255
- [Background] Agarwala P, Salzman SH. Six-Minute Walk Test: Clinical Role, Technique, Coding, and Reimbursement. Chest. 2020 Mar;157(3):603-611. doi: 10.1016/j.chest.2019.10.014. Epub 2019 Nov 2. PMID 31689414
- [Background] Ceron C, Otto D, Signorini AV, Beck MC, Camilis M, Sganzerla D, Rosa RG, Teixeira C. The Effect of Speaking Valves on ICU Mobility of Individuals With Tracheostomy. Respir Care. 2020 Feb;65(2):144-149. doi: 10.4187/respcare.06768. Epub 2019 Oct 15. PMID 31615923
- See also: Borg Rating of Perceived Exertion; Physio-Pedia — https://www.physio-pedia.com/Borg_Rating_Of_Perceived_Exertion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited from the inpatient population admitted to Gaylord Hospital.
Pre-assignment Details: Patients were excluded from study inclusion if they did not meet one or more study criteria.
Period: Overall Study
Arm/Group | Speaking Valve, Then Open Tracheostomy | Open Tracheostomy, Then Speaking Valve
Started | 13 | 13
Completed | 11 | 13
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Tracheostomy, Then Speaking Valve | Speaking Valve, Then Open Tracheostomy | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants] — Age at time of study consent and enrollment is reported.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 7 | 12
    >=65 years | 8 | 6 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 10 | 6 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Six Minute Walk Test - First Paired Sessions
Description: During each session, Participants will be asked to walk as far as possible along a corridor for a period of six minutes. The distance the Participant walks will be recorded to compare if the Participant can walk further with or without the PMV in place. Participant can use a device to assist with balance and the Participant can be assisted by an investigator, if needed. Each session is scheduled in an alternating fashion for whether or not Participant will use the PMV (i.e. day one no PMV, day two with PMV, day three no PMV, day four with PMV). Participants will complete 3 sessions with the PMV in place and 3 sessions with an open tracheostomy. Study sessions will occur on consecutive days, five days a week, Monday through Friday, until a minimum of 2 to maximum of 6 sessions are completed. This will equate to 1 to 3 completed paired sessions.
Time Frame: The first paired study session (Day 1) will occur within 72 hours of the participant being cleared by Medical Staff for PMV use. The second paired session will occur the day after session 1 (Day 2).
Population: Ambulation distance (feet)
Measure: Mean (Standard Deviation); unit: Feet
Groups:
- Speaking Valve: Speaking valve in place: Participants will perform the six minute walk test with a PMV in place. Participants will complete 1 to 3 sessions over approximately three-weeks.
Arm/Group | Speaking Valve | Open Tracheostomy
Number analyzed (Participants) | 24 | 24
Feet | 413 (348) | 387 (301.1)
Statistical Analysis 1: Comparison: Speaking Valve vs Open Tracheostomy; Test type: Superiority; p = 0.2795, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -26.08, 95% CI 2-sided [-74.80 to 22.63]

2. Primary Outcome: Six Minute Walk Test - Second Paired Sessions
Description: as for outcome 1
Time Frame: The third study session (Day 3) will occur the day following the second study session (Day 2). The fourth study session (Day 4) will occur the day following the third study session (Day 3).
Population: Complete paired datasets from sessions 3-4. This number may be less than the overall recruitment number due to discharge from hospital or study drop-out.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Speaking Valve | Open Tracheostomy
Number analyzed (Participants) | 5 | 5
Feet | 350 (378.81) | 384.6 (386.61)

3. Primary Outcome: Six Minute Walk Test - Third Paired Sessions
Description: as for outcome 1
Time Frame: The fifth study session (Day 5) will occur the day following the fourth study session (Day 4). The sixth study session (Day 6) will occur the day following the fifth study session (Day 5).
Population: Complete paired datasets from sessions 5-6. This number may be less than the overall recruitment number due to discharge from hospital or study drop-out.
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Speaking Valve | Open Tracheostomy
Number analyzed (Participants) | 2 | 2
Feet | 380 (84.85) | 357.5 (166.17)

4. Primary Outcome: Average Change of Borg Rating of Perceived Exertion - First Paired Sessions
Description: Borg Rating of Perceived Exertion is a self reported outcome score, based on a scale of 6 through 20 (20 being the hardest or most exertion, 6 being the least exertion).
  The first session will occur within 72 hours of the participant being cleared by Medical Staff for PMV use. Subsequent sessions will occur on every consecutive day following for 6 days total, Monday through Friday, until a minimum of 2 to maximum of 6 sessions are completed. This will equal 1 to 3 paired sessions. Average change will be calculated by using Post intervention scores subtracted by Pre intervention scores.
Time Frame: as for outcome 1
Population: BORG change from before session to after session
Measure: Mean (Standard Deviation); unit: Change of score on a scale
Arm/Group | Speaking Valve | Open Tracheostomy
Number analyzed (Participants) | 23 | 23
Change of score on a scale | 4.35 (2.92) | 3.65 (2.52)
Statistical Analysis 1: Comparison: Speaking Valve vs Open Tracheostomy; Test type: Superiority; p = 0.3416, t-test, 2 sided; Paired t-test; Mean Difference (Final Values) = -0.6957, 95% CI 2-sided [-2.179 to 0.7877]

5. Primary Outcome: Average Change of Borg Rating of Perceived Exertion - Second Paired Sessions
Description: as for outcome 4
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change of score on a scale
Arm/Group | Speaking Valve | Open Tracheostomy
Number analyzed (Participants) | 5 | 5
Change of score on a scale | 6 (4.06) | 5.8 (4.82)

6. Primary Outcome: Average Change of Borg Rating of Perceived Exertion - Third Paired Sessions
Description: as for outcome 4
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Change of score on a scale
Arm/Group | Speaking Valve | Open Tracheostomy
Number analyzed (Participants) | 2 | 2
Change of score on a scale | 4.5 (0.71) | 8 (1.41)

7. Secondary Outcome: Change in Heart Rate - First Paired Sessions
Description: Using a finger pulse-oxygen meter. These are paired data from session 1 and session 2. Change will be calculated using Post intervention scores minus Pre intervention scores.
Time Frame: Participant heart rate will be measured just prior and immediately after each intervention.
Population: Heart rate (BPM) change from before session to after session
Measure: Mean (Standard Deviation); unit: Change in beats per minute
Arm/Group | Speaking Valve | Open Tracheostomy
Number analyzed (Participants) | 24 | 24
Change in beats per minute | 18 (12.5) | 15.4 (12.4)

8. Secondary Outcome: Change in Oxygen Saturation - First Paired Sessions
Description: as for outcome 7
Time Frame: Participant oxygen saturation will be measured just prior and immediately after each intervention.
Population: Oxygen Saturation (%) change from before session to after session
Measure: Mean (Standard Deviation); unit: Change in O2 Saturation percentage
Arm/Group | Speaking Valve | Open Tracheostomy
Number analyzed (Participants) | 24 | 24
Change in O2 Saturation percentage | -3.6 (4.3) | -2.3 (3.9)

9. Secondary Outcome: Active Standing Time - First Paired Sessions
Description: The duration of active standing time, including standing rest breaks and active ambulation, that participants are able to tolerate while completing the six-minute walk test will be recorded. These are paired data from session 1 and session 2.
Time Frame: Participant active standing time will be recorded immediately after each intervention.
Population: Time (Seconds)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Speaking Valve | Open Tracheostomy
Number analyzed (Participants) | 24 | 24
seconds | 259 (110) | 257 (113)

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events during the course of enrollment in study activities, on average 1 month from baseline.
Description: The definition of adverse event and/or serious adverse event did not differs from the clinicaltrials.gov definition.
Arm/Group | Speaking Valve | Open Tracheostomy
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT04941456/Prot_SAP_000.pdf